CLINICAL TRIAL: NCT04770116
Title: The Effect of Sleep and Slow Wave Enhancement on Recovery From a Concussion in Children and Adolescents: A Longitudinal, Randomized, Double-Blind, and Sham-Controlled Study
Brief Title: Auditory Slow Wave Enhancement After Concussion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: ETH Zurich (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-00253
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Concussion Post Syndrome
Keywords: sleep; auditory stimulation; post-concussive symptoms; in-home EEG
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study helpers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group will receive all-night auditory stimulation during sleep over one week using a portable, in-home device (MHSL-SleepBand).
  Interventions: Device: Auditory Stimulation
- Control group (Sham Comparator): Participants in this group will receive sham-stimulation, i.e. the device will be applied (biosignals will be recorded), but no tones will be played.
  Interventions: Device: Auditory Stimulation

INTERVENTIONS:
Device: Auditory Stimulation — The device records biosignals and precisely plays tones to enhance sleep slow waves.

SUMMARY:
The prevalence of a traumatic brain injury (TBI) in children and adolescents is around 30% with 70-90% being classified as mild (concussion). Because the brain of a child is still developing, a TBI can have devastating effects and possibly creates lifetime challenges. Sleep seems to play an important role in the post-concussion recovery process. Auditory stimulation during sleep has been shown to reliably boost slow waves, a solid marker for the depth of sleep, and can thus be used to deepen sleep. This study aims to investigate the effects of sleep enhancement via auditory stimulation on recovery after a concussion in children and adolescents in their home. Therefore, half of the patients receive one week of auditory stimulation during deep sleep at their home using a mobile device. The other half follows the same study protocol, but no tones are administered (sham). Cognitive tests as well as symptom questionnaires are used to assess the recovery process. It is hypothesized that the patients in the intervention group will recover better than the ones who haven't received the intervention. Additionally, a group of children and adolescents who never sustained a concussion is included as a control.

DETAILED DESCRIPTION:
In total, 120 participants are planned: 60 patients (30 intervention, 30 sham) and 60 controls (30 intervention, 30 sham). This was estimated from a power analysis and based on previous results. Patients are recruited from the University Children's Hospital Zurich.

At first, the participants will complete a baseline assessment of neuropsychological measures (cognitive tests and questionnaires). After completion of the baseline assessment, the participants receive deep sleep enhancement with auditory stimulation for seven nights, but half of them will only receive sham stimulation (device application, but no stimulation). Additionally, they wear an actigraph throughout the whole week. Afterwards, they fill in again some questionnaires (intermediate assessment). One month after study inclusion, the first follow-up will take place where neuropsychological and (optionally) neurological measures will be collected. The second follow-up takes place six months after study inclusion and involves again filling in questionnaires about post-concussive symptoms.

The study will be monitored regularly in terms of data validation and source data verification. Adverse events and device deficiencies are carefully documented and reported according to the guidelines of swissmedic and the responsible ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age between 6 and 18 years
* Good knowledge of German of the patient and at least one legal representative
* Patients: Presentation to the Emergency of the University Children's Hospital Zurich because of a concussion (diagnosed by medical doctor)

Exclusion Criteria:

* Preterm birth (< 37 gestational weeks)
* Diagnosed hearing disorder
* Psychiatric, syndromal, or neurological pre-existing condition (except for previous concussion)
* Skin disorder/skin problem in the face/ear area that requires Treatment
* Usage of neuroactive substances
* Patients: Concomitant injury that requires intense pain medication or a prolonged hospital stay, or that causes limited use of the dominant Hand
* Patients: Previous moderate-severe TBI
* Controls: Injury of the dominant hand, on head, arm, or leg
* Controls: Previous TBI (of any severity)

Additional inclusion criteria for the optional MRI measurement for both groups:

* Age at least 8 years
* Fulfilment of all MRI safety criteria
* The participant and the legal representative would want to know about incidental findings.
* Girls: No pregnancy or breast feeding.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance - attention | Measured one month after study inclusion.
  Assessed by standardized test (normative values).
Cognitive Performance - processing speed | Measured one month after study inclusion.
  Assessed by standardized test (normative values).
Cognitive Performance - executive function | Measured one month after study inclusion.
  Assessed by standardized test (normative values).

SECONDARY OUTCOMES:
Subjective recovery | Measured at baseline, one week later (intermediate assessment), one month later (follow-up 1) and six months later (follow-up 2).
  Assessed by standardized symptom questionnaires.
Algorithm performance | Recorded during seven nights of stimulation or sham (intervention week).
  The algorithm flags which are produced by the mobile device used for the auditory stimulation (i.e. sleep detection flags, stimulation flags). They are used to investigate the algorithm performance for each subject.
Neurological outcome | One month after study inclusion (follow-up 1).
  Measured using Magnetic Resonance Imaging (standard structural and hemodynamic imaging, DTI, and susceptibility weighting) to investigate the neurological outcome.
Injury characteristics | baseline, pre-intervention
  Only for patients: Injury characteristics collected from the Hospital Information System that might influence baseline and follow-up measures and their change over time.
Other possible moderators of the Intervention | Collected at the baseline assessment.
  For example age and socio-economic status.
EEG power | Recorded during the intervention week.
  Power in frequency bands (delta, theta, alpha, beta, gramma).
Sleep stages | Recorded during the intervention week.
  EEG, EOG and EMG used for sleep scoring (sleep stages).
Sleep EEG characteristics | Recorded during the intervention week.
  Characteristics of sleep EEG Features (slow waves, spindles).
Subjective sleep | Collected throughout the whole study participation, in total 6 months (baseline, one week later (intermediate assessment), one month later (follow-up 1) and six months later (follow-up 2)).
  Assessed by standardized questionnaire
Actigraphy | Recorded during the intervention week.
  Measured by GENEActiv (activity bouts).
Objective and subjective sleep measures | Recorded at all study visits over a period of six months (baseline assessment, intervention week, follow-up 1 and follow-up 2)..
  Sleep measured by EEG and actigraphy (objective) as well as questionnaires (subjective)

OTHER OUTCOMES:
Intervention tolerability | After the intervention week (one week after study inclusion).
  Measured using an intervention evaluation questionnaire (self-designed).

CONTACTS AND LOCATIONS:
Overall Officials: Reto Huber, Prof., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland